CLINICAL TRIAL: NCT05908058
Title: The Investigation of Emotional Changes Between Emergency and Intensive Care Unit and On-site Counter Staffs After COVID-19 Infection and Exploring The Impact of Personnel Emotional Adjustment About Duty and Future Planning
Brief Title: Emotional Changes Between Emergency and Intensive Care Unit and On-site Counter Staffs After COVID-19 Infection
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: St. Martin De Porress Hospital (Other)
Responsible Party: Principal Investigator, Chia-hsi Chen, doctor, St. Martin De Porress Hospital
Other Study IDs: 23B-003
Record Dates: First submitted 2023-06-15; First posted 2023-06-18 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Psychological Distress; COVID-19 Infection; Anxiety and Fear-Related Disorders
Keywords: Emotional Change; COVID-19 Infection; Personnel Emotional Adjustment; Duty and Future Planning
MeSH Terms: conditions — COVID-19; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Emotional Changes Investigation — Emotional Changes between Emergency and Intensive care unit and On-site Counter Staffs after COVID-19 Infection and Exploring The Impact of Personnel Emotional Adjustment

SUMMARY:
The emotional and work changes of the staffs and the on-site counter staffs will have a certain impact during this pandemic period. Because a large number of critically ill patients are obstructive in emergency and critical care uint. It will induce a huge impact on the deployment of medical team manpower The purpose of this study is to understand the situation of emergency and intensive care unit personnel after covid-19 infection. It will help the hospital superintendent to understand the impact of emotional adjustment on its own work, understand the emotional situation of on-site personnel, future planning and r deployment.

DETAILED DESCRIPTION:
The emotional and work changes of the staffs and on-site counter staffs will have a certain impact during this pandemic period. Because a large number of critically ill patients are obstructive in emergency and critical care unit. It will induce a huge impact on the deployment of medical team manpower The purpose of this study is to understand the situation of emergency and intensive care unit personnel after COVID-19 infection. It will help the hospital superintendent to understand the impact of emotional adjustment on its own work, understand the emotional situation of on-site personnel, future planning and r deployment.

1. Explore the emotional changes of on-site emergency department and critical care unit staffs and on-site counter staffs by filling in questionnaires
2. Understand the emotional changes of personnel in various units and on-site counter personnel and how to adjust.
3. Arrange the Likert scale questionnaire with Meleis Nursing Transitional Theory. The different aspects of the questionnaire to quantify the emotional changes of the emergency and critical unit personnel and the on-site counter personnel. Each questionnaire takes about 20 minutes to 30 minutes to fill this questionnaire.
4. Analyze the emotional adjustment of the staffs in the acute and severe unit that affects their own work and how to affect the relationship between colleagues and medical practice execution.
5. This study uses empirical evidence to analyze and evaluate the emotional changes of emergency department and intensive care unit personnel and on-site counter personnel, understand the rationality of hospital manpower deployment and make the assistance needed

ELIGIBILITY:
Inclusion Criteria:

* emergency department and intensive care unit personnel after facing their own infection with COVID-19.

Exclusion Criteria:

* Exclude those who fill in the questionnaire with incomplete information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: emergency department and intensive care unit staffs with COVID 19 infection
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
The Investigation of Emotional Changes between Emergency and Intensive care unit and On-site Counter Staffs after COVID-19 Infection and Exploring The Impact of Personnel Emotional Adjustment about Duty and Future Planning | 2 months
  There is a huge impact on the deployment of medical team manpower after critically ill patients accumulated in emergency room and critical care unit. The purpose of this study is to understand the emotional change situation of emergency and intensive care unit personnel after covid-19 infection.
  It will help the superintendent to understand the impact of emotional adjustment on its own work, understand the situation of on-site personnel and adjust manpower planning and deployment.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsi Chen, Dr, Principal Investigator — St. Martin De Porres Hospital, Emergency Medicine Department
Locations (1):
- St. Martin De Porres Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be held by Dr principal investigator and no data sharing is necessary.

REFERENCES:
- [Result] Aydin R, Bulut E. Experiences of nurses diagnosed with COVID-19 in Turkey: A qualitative study. Int Nurs Rev. 2022 Sep;69(3):294-304. doi: 10.1111/inr.12735. Epub 2021 Dec 18. PMID 34921729
- See also: A qualitative study in Turkey about the experiences of nurses diagnosed with COVID-19 A qualitative study in Turkey — http://pubmed.ncbi.nlm.nih.gov/34921729/